CLINICAL TRIAL: NCT04630613
Title: NOX4, Mitochondria and Related Biomarkers in Autosomal Dominant Polycystic Kidney Disease
Brief Title: NOX4 and Related Biomarkers in ADPKD
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Polycystic Kidney Disease Foundation (Other)
Responsible Party: Principal Investigator, Maria V. Irazabal Mira, Principal Investigator, Mayo Clinic
Other Study IDs: 18-000637
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Oxidative Stress; Mitochondria injury and function; NADPH oxidase 4
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Urine and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a previous diagnosis of ADPKD: Patients that have been diagnosed with ADPKD and are classified as Class 1A, 1B, 1C, 1D and 1E.

SUMMARY:
To determine the value of NOX4, markers of mitochondria injury and function, and oxidative stress as real-time biomarkers to assess disease severity in patients with early autosomal dominant polycystic kidney disease (ADPKD).

DETAILED DESCRIPTION:
This will be a cross sectional study and will include male and female, young (15-40-years) well characterized patients with early (eGFR>70mL/min/1.73m2) ADPKD. Patients with different classes of disease severity will be selected using the ADPKD imaging classification. The study will include 60 class-1 (A-E) patients (N=12 per each sub-class).

ELIGIBILITY:
Inclusion Criteria:

* ADPKD (based on Ravine et al. criteria)
* Class 1 A-E according to imaging classification
* Male and female subjects 15 - 40 years of age
* Estimated GFR> 70 mL/min/1.73 m2 (CKD-EPI)
* Ability to provide written, informed consent

Exclusion Criteria:

* Class 2 according to imaging classification
* Concomitant systemic disease affecting the kidney
* Diabetes mellitus
* Predicted urine protein excretion in >1 g/24 hrs
* Use of antioxidants i.e. vitamins, Nrf2 activators
* Abnormal urinalysis

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female patients with a previous diagnosis of ADPKD
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
NOX4 levels | Baseline
  Determination of NOX4 levels from urine and plasma samples
mtDNA copy number | Baseline
  Determination of mtDNA copy number from urine and plasma samples
Tricarboxylic Acid (TCA) cycle metabolites | Baseline
  Determination of TCA cycle metabolite concentration from urine and plasma samples
REDOX status | Baseline
  Determination of REDOX from urine and plasma samples
Total kidney volume (TKV) | Baseline
  Determined by MRI

SECONDARY OUTCOMES:
Estimated Glomerular Filtration Rate (eGFR) | Baseline
  Estimated by CKD-epi equation

CONTACTS AND LOCATIONS:
Overall Officials: Maria V Irazabal, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials